CLINICAL TRIAL: NCT06442540
Title: Effects of Intra Muscular Electrotherapy Combined With Manipulative Therapy in Patients With Sacral Torsion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/11
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): HVLA thrust for SI Joint once per week:
  Core stability exercises Intramuscular electrotherapy / 3 sessions per week 10 mins / frequency 100hz muscles( piriformis, erector spinae )
  Interventions: Procedure: Manipulation; Procedure: Core Stability Exercises; Procedure: Intramusular electrotherapy
- Group 2 (Experimental): Hot pack 10 mins soft tissue / myofacial release ( piriformis, erector spinae ) Piriformis stretching core stability exercises
  Interventions: Procedure: Physical Agents; Procedure: Core Stability Exercises; Procedure: Soft tissue mobility

INTERVENTIONS:
Procedure: Physical Agents — Hot pack
  Arms: Group 2
Procedure: Manipulation — HVLA manipulation of SI joint
  Arms: Group 1
Procedure: Core Stability Exercises — Supine abdominal draw-in Hold 8s 3s off x 2 Abdominal draw-in, with one knee drawn to the chest. Hold 8s 3s off x 2 Abdominal draw-in, with the heels sliding backward one after the other. 10 reps 3s off x 2 Abdominal draw-in, with both knees drawn to the chest. Hold 8s 3s off x 2 Supine twist 15 reps 3s off x 3 Prone bridging on elbows Hold 8s 3s off x 3 Side bridging on elbows Hold 8s 3s off x 3 Quadruped opposite arm-leg lift Hold 8s 3s off x 3 Advance to the stage 2 when the patient can hold 30 reps for an 8-sec hold.
Procedure: Intramusular electrotherapy — Intramuscular electrotherapy/ 3 sessions per week
  Arms: Group 1
Procedure: Soft tissue mobility — Stretching and Myofacial Release of piriformis and erector spinae
  Arms: Group 2

SUMMARY:
This study is a randomised controlled trial and the purpose of this study is to determine the effect of intra muscular electrotherapy combined with manipulative therapy in terms of pain, mobility, range of motion, and disability."

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of intra muscular electrotherapy combined with manipulative therapy in terms of pain, mobility, range of motion, and disability in patients with sacral torsion." (age : 22-44 years )

1. Numeric pain rating scale
2. Inclinometer Lumbar Flexion
3. Oswestry Disability Questionairre
4. Goniometer SLR ROM Data will be collected before and after the intervention protocol for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Age group: 22-44 years old
* Both males and females
* Clinically diagnosed sacral torsion
* Patients with pain intensity of at least 5 on NPRS
* Positive backward bent test
* Positive forward bent test
* Uneven Sacral sulcus
* Uneven ILA of sacrum
* Piriformis syndrome

Exclusion criteria :

* Any congenital deformities
* Demonstrated neurological deficit.
* Pregnant females
* History of spinal surgery
* Spondylolisthesis
* Severe lumbar spondylosis
* Spinal stenosis
* Serious spinal conditions like infection, tumors, osteoporosis, spinal fracture
* osteoporosis

Ages: 22 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  Numeric Pain Rating Scale (NPRS): ICC (0.93-0.96) It has a scale of 0-10 or 0-100 points and can be given verbally or in writing
Lumbar ROM | 4 weeks
  Lumbar ROM will be measured using Inclinometer
SLR ROM | 4 weeks
  SLR ROM will be measured using Goniometer
Level of Disability | 4 Weeks
  Oswestry disability questionairre

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan